CLINICAL TRIAL: NCT04332653
Title: An Open-label Phase 1b/2a Study of NT-I7 (Efineptakin Alfa) in Combination With Pembrolizumab in Subjects With Relapsed/Refractory Advanced Solid Tumors
Brief Title: NT-I7 (Efineptakin Alfa) in Combination With Pembrolizumab in Participants With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NeoImmuneTech (Industry)
Collaborators: Merck Sharp and Dohme LLC, Rahway, NJ, USA (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NIT-110; MK-3475-A60 (Other: Merck Sharp and Dohme LLC, Rahway, NJ, USA); KEYNOTE-A60 (Other: Merck Sharp and Dohme LLC, Rahway, NJ, USA)
Record Dates: First submitted 2020-03-31; First posted 2020-04-03 (Actual); Results first posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Any Advanced Solid Tumors; Triple Negative Breast Cancer; Non Small Cell Lung Cancer; Small Cell Lung Cancer; Microsatellite Stable Colorectal Cancer; Pancreatic Cancer; Ovarian Cancer
Keywords: NT-I7 (Efineptakin alfa); Solid Tumor; Pembrolizumab; Neoplasms; Lung; Breast; Pancreas; Colorectal; Non-small Cell Lung; Small Cell Lung; Thoracic Neoplasms; Interleukin 7; Carcinoma; Cancer; Programmed cell death protein (PD-1); Ovarian
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Pancreatic Neoplasms; Ovarian Neoplasms; Neoplasms; Thoracic Neoplasms; Carcinoma; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — efineptakin alfa; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Phase 1b: NT-I7 Dose Escalation (Experimental): NT-I7 will be administered on Day 1 of alternate 21 day cycles (Cycle 1, 3, 5 etc.). Dosage will increase until the maximum tolerated dose (MTD) and/or the recommended phase 2 (RP2D) dose is reached.
  Pembrolizumab will be administered on Day 1 of every 21 day cycle.
  Interventions: Drug: NT-I7; Drug: pembrolizumab (KEYTRUDA®)
- Phase 2a: CPI Treated Triple Negative Breast Cancer (Experimental): Participants with checkpoint inhibitor (CPI) treated relapsed or refractory triple negative breast cancer (TNBC). Participants will receive the recommended phase 2 dose (RP2D) identified during Phase 1b.
  Pembrolizumab will be administered on Day 1 of every 21 day cycle.
  Interventions: Drug: NT-I7; Drug: pembrolizumab (KEYTRUDA®)
- Phase 2a: CPI Treated Non-small Cell Lung Cancer (Experimental): Participants with checkpoint inhibitor (CPI) treated relapsed or refractory non-small cell lung cancer (NSCLC). Participants will receive the recommended phase 2 dose (RP2D) identified during Phase 1b.
  Pembrolizumab will be administered on Day 1 of every 21 day cycle.
  Interventions: Drug: NT-I7; Drug: pembrolizumab (KEYTRUDA®)
- Phase 2a: CPI Treated Small Cell Lung Cancer (Experimental): Participants with checkpoint inhibitor (CPI) treated relapsed or refractory small cell lung cancer (SCLC). Participants will receive the recommended phase 2 dose (RP2D) identified during Phase 1b.
  Pembrolizumab will be administered on Day 1 of every 21 day cycle.
  Interventions: Drug: NT-I7; Drug: pembrolizumab (KEYTRUDA®)
- Phase 2a: CPI Naïve Microsatellite Stable Colorectal Cancer (Experimental): Participants with checkpoint inhibitor (CPI) naïve relapsed or refractory microsatellite stable colorectal cancer (MSS-CRC). Participants will receive the recommended phase 2 dose (RP2D) identified during Phase 1b.
  Pembrolizumab will be administered on Day 1 of every 21 day cycle.
  Interventions: Drug: NT-I7; Drug: pembrolizumab (KEYTRUDA®)
- Phase 2a: CPI Naïve Pancreatic Cancer (Experimental): Participants with checkpoint inhibitor (CPI) naïve relapsed or refractory pancreatic cancer (PC). Participants will receive the recommended phase 2 dose (RP2D) identified during Phase 1b.
  Pembrolizumab will be administered on Day 1 of every 21 day cycle.
  Interventions: Drug: NT-I7; Drug: pembrolizumab (KEYTRUDA®)
- Phase 2a: CPI Naïve Microsatellite Stable Colorectal Cancer, Expansion Cohort (Experimental): Participants with checkpoint inhibitor (CPI) naïve relapsed or refractory microsatellite stable colorectal cancer (MSS-CRC). Participants will receive 1200 µg/kg of NT-I7 and and a fixed dose of 200 mg of pemprolizumab.
  Pembrolizumab will be administered on Day 1 of every 21 day cycle.
  Interventions: Drug: NT-I7; Drug: pembrolizumab (KEYTRUDA®)
- Phase 2a: CPI Naïve Pancreatic Cancer, Expansion Cohort (Experimental): Participants with checkpoint inhibitor (CPI) naïve relapsed or refractory pancreatic cancer (PC).Participants will receive 1200 µg/kg of NT-I7 and a fixed dose of 200 mg of pemprolizumab.
  Pembrolizumab will be administered on Day 1 of every 21 day cycle.
  Interventions: Drug: NT-I7; Drug: pembrolizumab (KEYTRUDA®)
- Biomarker Cohort: CPI Naïve Ovarian Cancer (Experimental): Participants with checkpoint inhibitor (CPI) naïve relapsed or refractory ovarian cancer (OC). Participants will receive a starting dose of 960 µg/kg of NT-I7 and a fixed dose of 200 mg of pemprolizumab.
  Pembrolizumab will be administered on Day 1 of every 21 day cycle.
  Interventions: Drug: NT-I7; Drug: pembrolizumab (KEYTRUDA®)

INTERVENTIONS:
Drug: NT-I7 — Administered by intramuscular (IM) injection
  Other Names: Efineptakin alfa; rhIL-7-hyFc
Drug: pembrolizumab (KEYTRUDA®) — Administered by intravenous (IV) injection
  Other Names: KEYTRUDA®

SUMMARY:
The main purposes of Phase 1b of this study are to determine the following in participants with advanced solid tumors:

* Safety and tolerability of NT-I7 in combination with pembrolizumab
* Maximum Tolerated Dose (MTD) and/or the Recommended Phase 2 Dose (RP2D)

The main purpose of Phase 2a of this study is to assess the preliminary anti-tumor activity of NT-I7 in combination with pembrolizumab in participants with checkpoint inhibitor (CPI) treated and naïve relapsed and refractory (R/R) tumors.

The main purpose of the Biomarker Cohort is to assess a potential correlation between tumor infiltrating lymphocytes (TILs) and clinical benefits in participants with CPI-naïve R/R ovarian cancer (OC).

DETAILED DESCRIPTION:
This is a multicenter, open-label Phase 1b/2a study of NT-I7 in combination with pembrolizumab. The study consists of a dose escalation phase (Phase 1b) followed by a dose expansion phase (Phase 2a) and a Biomarker Cohort.

The Phase 1b is designed to assess the safety and tolerability, including determination of the Maximum Tolerated Dose (MTD) and/or the Recommended Phase 2 Dose (RP2D) of NT-I7.

The main purpose of Phase 2a of this study is to assess the preliminary antitumor activity of NT-I7 in combination with pembrolizumab in participants with relapsed/refractory

* checkpoint inhibitor (CPI)-treated Triple Negative Breast Cancer (TNBC), Non-small Cell Lung Cancer (NSCLC), and Small Cell Lung Cancer (SCLC)
* checkpoint inhibitor (CPI)-naïve Microsatellite Stable Colorectal Cancer (MSS-CRC), and Pancreatic Cancer (PC) The Biomarker Cohort is designed to assess the correlation between tumor infiltrating lymphocytes (TILs) and clinical benefits of NT-I7 in combination with pembrolizumab in participants with CPI naïve R/R Ovarian Cancer (OC).

ELIGIBILITY:
Inclusion Criteria:

(Participants must meet all the following to be eligible)

* Participants with histologically or cytologically confirmed advanced or metastatic solid tumors.
* Have measurable disease per RECIST v1.1.
* Participants enrolling in the Phase 1b, Arms I, IV, IVa, V, and Va of the Phase 2a, and the Biomarker Cohort OC must have biopsiable disease.
* Female participants who are either postmenopausal for at least 1 year, are surgically sterile for at least 6 weeks; female participants of childbearing potential must agree to remain abstinent (refrain from heterosexual intercourse) or to use dual methods of contraception for the duration of study treatment and for 120 days after the last dose of study treatment (pembrolizumab and/or NT-I7).
* Non-sterile male participants who are sexually active with female partners of childbearing potential must agree to remain abstinent (refrain from heterosexual intercourse) or to use highly effective method(s) of contraception for the duration of study treatment and for 120 days after the last dose of study treatment (pembrolizumab and/or NT-I7).
* Meet the requirements for the intended stages and arms (disease specific inclusion criteria), as follows:

Applicable to the Dose escalation phase (Phase 1b) only: (Biopsy Arm)

* Relapsed/refractory advanced solid tumors.

Applicable to the Dose expansion phase (Phase 2a) only:

Anti-PD-1/anti-PD-L1 refractory criteria for CPI-treated TNBC, NSCLC, and SCLC

* Has received at least 2 doses of an approved anti-PD-1/anti-PD-L1 monoclonal antibody (mAb).
* Has demonstrated disease progression after anti-PD-1/anti-PD-L1.

Specific to Arm I: CPI-treated R/R TNBC (Biopsy Arm)

* Histopathologic or cytologic documented TNBC.
* Received one or more prior therapies for TNBC in the advanced or metastatic setting, and prior treatment (for advanced, metastatic or (neo) adjuvant).

Specific to Arm II: CPI-treated R/R NSCLC

* Had prior treatment with CPI. Participants with estimated glomerular filtration rate (EGFR), BRAF, or c-ros oncogene 1(ROS1) mutations or anaplastic lymphoma kinase (ALK) translocations are required to have received prior therapy with the appropriate tyrosine kinase inhibitor (TKI).

Specific to Arm III: CPI-treated R/R SCLC

* Recurrent extensive-stage SCLC; Received prior CPI therapy.

Specific to Arm IV and IVa: CPI-naïve R/R MSS-CRC (Biopsy Arm)

* MSS-CRC (categorized as MSS by immunohistochemistry(IHC) or polymerase chain reaction (PCR).
* Previously treated with standard therapies, which must include fluoropyrimidine, oxaliplatin, and irinotecan; participants treated with CPI are not eligible.

Specific to Arm V and Va: CPI-naïve R/R Pancreatic Cancer (Biopsy Arm)

* Have documented radiographic progression to or documented in tolerance of first line systemic chemotherapy which included either gemcitabine or Fluorouracil (5-FU)-based regimen (including capecitabine); participants treated previously with CPI are not eligible.

Specific to Biomarker Cohort: CPI-naïve R/R Ovarian Cancer

* Up to 5 prior lines of treatment, including platinum-based treatment(s); participants treated previously with CPIs are not eligible.
* Willing to provide pre- and on-treatment tumor biopsies.

Exclusion Criteria:

* Pregnant, lactating or breastfeeding.
* Receiving chemotherapy or any anti-cancer therapy (approved or investigational) with half-life <1 week within 30 days or 5 half-lives.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate if stable.
* Participants who have received treatment with systemic immunosuppressive medications.
* Has a history of non-infectious pneumonitis that required steroids or current pneumonitis.
* Has had an allogenic tissue/solid organ transplant or bone marrow transplant.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX-40, CD137) and was discontinued from that treatment due to a Grade 3 or higher Immune related adverse event (irAE).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2020-06-10 (Actual); Primary Completion 2024-11-22 (Actual); Study Completion 2025-01-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Moffit Cancer Center, Tampa, Florida
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Mary Crowley Cancer Research, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 215 participants were enrolled in the United States from June 2020 to January 2025.
Pre-assignment Details: The trial consisted of a dose escalation phase (Phase 1b) followed by a dose expansion phase (Phase 2a) and a Biomarker Cohort.
Groups:
- Phase 1b: Dose Level 1 (NT-I7 480 ug/kg): Participants received NT-I7 as an intramuscular (IM) injection every 6 weeks (Q6W), on Day 1 of alternate cycles (Cycle 1, 3, 5 etc.). Participants received 200 mg Pembrolizumab as an intravenous (IV) infusion every 3 weeks (Q3W), on Day 1 of every cycle (cycle duration= 21 days).
- Phase 1b: Dose Level 2 (NT-I7 960 ug/kg); Phase 1b: Dose Level 3 (NT-I7 1200 ug/kg): Participants received NT-I7 as an IM injection Q6W, on Day 1 of alternate cycles (Cycle 1, 3, 5 etc.). Participants received 200 mg Pembrolizumab as an IV infusion Q3W, on Day 1 of every cycle (cycle duration= 21 days).
- Phase 2a: Arm I: Checkpoint inhibitor (CPI) treated participants with relapsed/refractory (R/R) triple negative breast cancer (TNBC) received NT-I7 at the recommended phase 2 dose (RP2D= 1200 ug/kg) as an IM injection Q6W, on Day 1 of alternate cycles (Cycle 1, 3, 5 etc.). Participants received 200 mg Pembrolizumab as an IV infusion Q3W, on Day 1 of every cycle (cycle duration= 21 days).
- Phase 2a: Arm II: CPI treated participants with R/R non-small cell lung cancer (NSCLC) received NT-I7 at the RP2D (1200 ug/kg) as an IM injection Q6W, on Day 1 of alternate cycles (Cycle 1, 3, 5 etc.). Participants received 200 mg Pembrolizumab as an IV infusion Q3W, on Day 1 of every cycle (cycle duration= 21 days).
- Phase 2a: Arm III: CPI treated participants with R/R small cell lung cancer (SCLC) received NT-I7 at the RP2D (1200 ug/kg) as an IM injection Q6W, on Day 1 of alternate cycles (Cycle 1, 3, 5 etc.). Participants received 200 mg Pembrolizumab as an IV infusion Q3W, on Day 1 of every cycle (cycle duration= 21 days).
- Phase 2a: Arm IV: CPI naïve participants with R/R microsatellite stable colorectal cancer (MSS-CRC) received NT-I7 at the RP2D (1200 ug/kg) as an IM injection Q6W, on Day 1 of alternate cycles (Cycle 1, 3, 5 etc.). Participants received 200 mg Pembrolizumab as an IV infusion Q3W, on Day 1 of every cycle (cycle duration= 21 days).
- Phase 2a: Arm IVa: Expansion Cohort. CPI naïve participants with R/R MSS-CRC received NT-I7 at the RP2D (1200 ug/kg) as an IM injection Q6W, on Day 1 of alternate cycles (Cycle 1, 3, 5 etc.). Participants received 200 mg Pembrolizumab as an IV infusion Q3W, on Day 1 of every cycle (cycle duration= 21 days).
- Phase 2a: Arm V: CPI naïve participants with R/R pancreatic cancer (PC) received NT-I7 at the RP2D (1200 ug/kg) as an IM injection Q6W, on Day 1 of alternate cycles (Cycle 1, 3, 5 etc.). Participants received 200 mg Pembrolizumab as an IV infusion Q3W, on Day 1 of every cycle (cycle duration= 21 days).
- Phase 2a: Arm Va: Expansion Cohort. CPI naïve participants with R/R PC received NT-I7 at the RP2D (1200 ug/kg) as an IM injection Q6W, on Day 1 of alternate cycles (Cycle 1, 3, 5 etc.). Participants received 200 mg Pembrolizumab as an IV infusion Q3W, on Day 1 of every cycle (cycle duration= 21 days).
- Phase 2a: Biomarker Cohort: CPI naïve participants with R/R ovarian cancer (OC) received NT-I7 960 ug/kg as an IM injection Q6W, on Day 1 of alternate cycles (Cycle 1, 3, 5 etc.). Participants received 200 mg Pembrolizumab as an IV infusion Q3W, on Day 1 of every cycle (cycle duration= 21 days).
Period: Phase 1b
Arm/Group | Phase 1b: Dose Level 1 (NT-I7 480 ug/kg) | Phase 1b: Dose Level 2 (NT-I7 960 ug/kg) | Phase 1b: Dose Level 3 (NT-I7 1200 ug/kg) | Phase 2a: Arm I | Phase 2a: Arm II | Phase 2a: Arm III | Phase 2a: Arm IV | Phase 2a: Arm IVa | Phase 2a: Arm V | Phase 2a: Arm Va | Phase 2a: Biomarker Cohort
Started | 3 | 3 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 2 | 3 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Progressive Disease | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase 2a
Arm/Group | Phase 1b: Dose Level 1 (NT-I7 480 ug/kg) | Phase 1b: Dose Level 2 (NT-I7 960 ug/kg) | Phase 1b: Dose Level 3 (NT-I7 1200 ug/kg) | Phase 2a: Arm I | Phase 2a: Arm II | Phase 2a: Arm III | Phase 2a: Arm IV | Phase 2a: Arm IVa | Phase 2a: Arm V | Phase 2a: Arm Va | Phase 2a: Biomarker Cohort
Started | 0 (Phase 1b and Phase 2a had separate populations.) | 0 (Phase 1b and Phase 2a had separate populations.) | 0 (Phase 1b and Phase 2a had separate populations.) | 16 (Phase 1b and Phase 2a had separate populations.) | 34 (Phase 1b and Phase 2a had separate populations.) | 17 (Phase 1b and Phase 2a had separate populations.) | 29 (Phase 1b and Phase 2a had separate populations.) | 28 (Phase 1b and Phase 2a had separate populations.) | 32 (Phase 1b and Phase 2a had separate populations.) | 34 (Phase 1b and Phase 2a had separate populations.) | 13 (Phase 1b and Phase 2a had separate populations.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not Completed | 0 | 0 | 0 | 16 | 34 | 17 | 29 | 28 | 32 | 34 | 12
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 9 | 20 | 12 | 18 | 16 | 18 | 24 | 8
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 1 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Progressive Disease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 3 | 0
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 3 | 1 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 4 | 11 | 5 | 9 | 5 | 11 | 4 | 3
Not completed — Miscellaneous | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase 1b: Dose Level 1 (NT-I7 480 ug/kg); Phase 1b: Dose Level 2 (NT-I7 960 ug/kg); Phase 1b: Dose Level 3 (NT-I7 1200 ug/kg): Participants received NT-I7 as an IM injection Q6W, on Day 1 of alternate cycles (Cycle 1, 3, 5 etc.). Participants received 200 mg Pembrolizumab as an IV infusion Q3W, on Day 1 of every cycle (cycle duration= 21 days).
- Phase 2a: Arm I: CPI treated participants with R/R TNBC received NT-I7 at the RP2D (1200 ug/kg) as an IM injection Q6W, on Day 1 of alternate cycles (Cycle 1, 3, 5 etc.). Participants received 200 mg Pembrolizumab as an IV infusion Q3W, on Day 1 of every cycle (cycle duration= 21 days).
- Phase 2a: Arm II: CPI treated participants with R/R NSCLC received NT-I7 at the RP2D (1200 ug/kg) as an IM injection Q6W, on Day 1 of alternate cycles (Cycle 1, 3, 5 etc.). Participants received 200 mg Pembrolizumab as an IV infusion Q3W, on Day 1 of every cycle (cycle duration= 21 days).
- Phase 2a: Arm III: CPI treated participants with R/R SCLC received NT-I7 at the RP2D (1200 ug/kg) as an IM injection Q6W, on Day 1 of alternate cycles (Cycle 1, 3, 5 etc.). Participants received 200 mg Pembrolizumab as an IV infusion Q3W, on Day 1 of every cycle (cycle duration= 21 days).
- Phase 2a: Arm IV: CPI naïve participants with R/R MSS-CRC received NT-I7 at the RP2D (1200 ug/kg) as an IM injection Q6W, on Day 1 of alternate cycles (Cycle 1, 3, 5 etc.). Participants received 200 mg Pembrolizumab as an IV infusion Q3W, on Day 1 of every cycle (cycle duration= 21 days).
- Phase 2a: Arm V: CPI naïve participants with R/R PC received NT-I7 at the RP2D (1200 ug/kg) as an IM injection Q6W, on Day 1 of alternate cycles (Cycle 1, 3, 5 etc.). Participants received 200 mg Pembrolizumab as an IV infusion Q3W, on Day 1 of every cycle (cycle duration= 21 days).
- Phase 2a: Biomarker Cohort: CPI naïve participants with R/R OC received NT-I7 960 ug/kg as an IM injection Q6W, on Day 1 of alternate cycles (Cycle 1, 3, 5 etc.). Participants received 200 mg Pembrolizumab as an IV infusion Q3W, on Day 1 of every cycle (cycle duration= 21 days).
- Total: Total of all reporting groups
Arm/Group | Phase 1b: Dose Level 1 (NT-I7 480 ug/kg) | Phase 1b: Dose Level 2 (NT-I7 960 ug/kg) | Phase 1b: Dose Level 3 (NT-I7 1200 ug/kg) | Phase 2a: Arm I | Phase 2a: Arm II | Phase 2a: Arm III | Phase 2a: Arm IV | Phase 2a: Arm IVa | Phase 2a: Arm V | Phase 2a: Arm Va | Phase 2a: Biomarker Cohort | Total
Number analyzed (Participants) | 3 | 3 | 6 | 16 | 34 | 17 | 29 | 28 | 32 | 34 | 13 | 215
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 5 | 12 | 15 | 8 | 26 | 21 | 15 | 16 | 8 | 131
  >=65 years | 0 | 1 | 1 | 4 | 19 | 9 | 3 | 7 | 17 | 18 | 5 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.0 (10.82) | 65.3 (10.12) | 54.8 (8.21) | 53.8 (10.75) | 65.2 (10.59) | 65.1 (6.85) | 54.7 (11.25) | 56.1 (10.37) | 65.1 (10.67) | 64.7 (9.49) | 58.1 (10.55) | 60.8 (11.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3 | 16 | 11 | 9 | 10 | 16 | 16 | 12 | 13 | 109
  Male | 2 | 1 | 3 | 0 | 23 | 8 | 19 | 12 | 16 | 22 | 0 | 106
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 2 | 0 | 0 | 2 | 3 | 2 | 3 | 0 | 14
  Not Hispanic or Latino | 2 | 2 | 4 | 14 | 31 | 17 | 25 | 24 | 29 | 30 | 13 | 191
  Unknown or Not Reported | 0 | 0 | 2 | 0 | 3 | 0 | 2 | 1 | 1 | 1 | 0 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 2 | 3 | 1 | 10
  Black or African American | 0 | 0 | 1 | 3 | 9 | 3 | 6 | 2 | 2 | 3 | 3 | 32
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  White | 2 | 1 | 3 | 11 | 23 | 13 | 22 | 22 | 27 | 25 | 9 | 158
  Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Not Reported | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 6
  Unknown | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 2 | 0 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 3 | 6 | 16 | 34 | 17 | 29 | 28 | 32 | 34 | 13 | 215

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b: Number of Participants Who Experienced Treatment Emergent Adverse Events (TEAEs), Serious AEs (SAEs), Trial Treatment-related TEAEs and Trial Treatment-related SAEs
Description: A TEAE was any AE that starts on/after the first day of trial treatment or that worsens on/after the first day of trial treatment and up to 30 days (90 days for serious adverse events) after the date of last dose of trial drugs, or initiation of new anticancer therapy, whichever is earlier. A SAE was defined as any AE that resulted in any of the following outcomes:
  1. Death;
  2. A life-threatening AE;
  3. An AE that resulted in inpatient hospitalization or prolongation of existing hospitalization for ≥24 hours;
  4. A persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions;
  5. A congenital anomaly/birth defect;
  6. Important Medical Events (IME) that may not result in death, be life threatening, or require hospitalization may be considered serious when, based upon medical judgment, they may jeopardize the participant and may require medical or surgical intervention to prevent one of the outcomes listed in this definition.
Time Frame: Up to 2 years and 3 months
Population: Safety Analysis Set: all participants who received at least one dose (even partially) of one or both trial medications. Only participants in Phase 1b were analyzed for this Outcome Measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Dose Level 1 (NT-I7 480 ug/kg) | Phase 1b: Dose Level 2 (NT-I7 960 ug/kg) | Phase 1b: Dose Level 3 (NT-I7 1200 ug/kg)
Number analyzed (Participants) | 3 | 3 | 6
Participants
  TEAEs | 3 | 3 | 6
  SAEs | 2 | 1 | 1
  Trial Treatment-related TEAEs | 3 | 2 | 6
  Trial Treatment-related SAEs | 1 | 0 | 0

2. Primary Outcome: Phase 1b: Number of Participants Who Experienced a Dose Limiting Toxicity (DLT)
Description: A DLT was defined as any AE occurring within the first 21 days that was considered to be related to the trial treatments (NT-I7 and/or pembrolizumab) per the investigator, and that met at least one of the non-hematologic or hematologic criteria:
  * Grade 4 non-hematologic toxicity
  * Grade ≥ 3 diarrhea, nausea and vomiting
  * Grade ≥ 3 rash for ≥ 5 days
  * Grade 4 neutropenia for ≥ 5 days
  * Febrile neutropenia Grade 3 or Grade 4
  * Other Grade 4 hematologic toxicity for ≥7 days, except thrombocytopenia
  * Any non-hematologic AE ≥ Grade 3 in severity
  * Any Grade 3 or Grade 4 non-hematologic laboratory value if medical intervention was required, led to hospitalization, persisted for > 1 week, resulted in potential drug-induced liver injury
  * Other Grade ≥ 3 clinical laboratory abnormalities not reversible to ≤ Grade 1 within 72 hours
  * Prolonged delay in initiating Cycle 2
  * Any treatment-related toxicity that caused treatment discontinuation in Cycle 1
  * Grade 5 toxicity.
Time Frame: Up to 21 days
Population: DLT Evaluable Analysis Set: all participants in Phase 1b portion of the study who were in safety analysis set and have completed the first 21 days (3 weeks) of study treatment (Cycle 1, Day 1 to 21) or any subjects who have not completed 21 days due to DLT.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Dose Level 1 (NT-I7 480 ug/kg) | Phase 1b: Dose Level 2 (NT-I7 960 ug/kg) | Phase 1b: Dose Level 3 (NT-I7 1200 ug/kg)
Number analyzed (Participants) | 3 | 3 | 6
Participants | 0 | 0 | 1

3. Primary Outcome: Phase 2a (Arms I to Va): Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants who had at least one confirmed partial response (PR) or complete response (CR), per Response Evaluation Criteria in Solid Tumors 1.1 (RECIST v1.1) and immune RECIST (iRECIST) as determined by the investigator. CR was defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have had reduction in short axis to <10 mm (<1 cm). PR was defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Up to 2 years
Population: Efficacy Evaluable Analysis Set: all participants who received at least one dose of both the trial medication (NT-I7 and Pembrolizumab) and had an evaluable baseline and at least one evaluable post-baseline assessment of tumor response. Only participants in Phase 2a (Arms I to Va) were analyzed for this Outcome Measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2a: Arm I | Phase 2a: Arm II | Phase 2a: Arm III | Phase 2a: Arm IV | Phase 2a: Arm IVa | Phase 2a: Arm V | Phase 2a: Arm Va
Number analyzed (Participants) | 14 | 26 | 15 | 27 | 26 | 26 | 26
percentage of participants
  ORR per RECIST 1.1 | 0 [0.0 to 23.2] | 0 [0.0 to 13.2] | 13.3 [1.7 to 40.5] | 3.7 [0.1 to 19.0] | 0 [0.0 to 13.2] | 3.8 [0.1 to 19.6] | 3.8 [0.1 to 19.6]
  ORR per iRECIST | 0 [0.0 to 23.2] | 3.8 [0.1 to 19.6] | 13.3 [1.7 to 40.5] | 11.1 [2.4 to 29.2] | 0 [0.0 to 13.2] | 7.7 [0.9 to 25.1] | 3.8 [0.1 to 19.6]

4. Primary Outcome: Biomarker Cohort: Percentage of Area Occupied by Tumor-Infiltrating Lymphocytes (TILs)
Description: CD8 positivity TILs in tumor biopsy samples were identified using a validated immunohistochemistry (IHC) assay and certified by a pathologist. The percentage of area occupied by TILs was evaluated in the stroma area, tumor area and tumor - relevant tissue area both pre- and post-treatment.
Time Frame: Pre-treatment and post-treatment (maximum duration of treatment of approximately 2 years)
Population: Safety Analysis Set: all participants who received at least one dose (even partially) of one or both trial medications. Only participants with positive CD8 marker were included.
Measure: Mean (Standard Deviation); unit: percentage of area occupied
Arm/Group | Phase 2a: Biomarker Cohort
Number analyzed (Participants) | 2
percentage of area occupied
  Stroma area: pre-treatment | 4.5 (4.95)
  Stroma area: post-treatment | 7.5 (3.54)
  Tumor area: pre-treatment | 0.5 (0.71)
  Tumor area: post-treatment | 0.5 (0.71)
  Tumor - relevant tissue area: pre-treatment | 4.5 (4.95)
  Tumor - relevant tissue area: post-treatment | 12.0 (11.31)

5. Secondary Outcome: Biomarker Cohort: ORR
Description: ORR was defined as the percentage of participants who had at least one confirmed PR or CR, per RECIST v1.1 and iRECIST as determined by the investigator. CR was defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have had reduction in short axis to <10 mm (<1 cm). PR was defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Up to 2 years
Population: Efficacy Evaluable Analysis Set: all participants who received at least one dose of both the trial medication (NT-I7 and Pembrolizumab) and had an evaluable baseline and at least one evaluable post-baseline assessment of tumor response. Only participants in Phase 2a (Biomarker Cohort) were analyzed for this Outcome Measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2a: Biomarker Cohort
Number analyzed (Participants) | 12
percentage of participants
  ORR per RECIST 1.1 | 16.7 [2.1 to 48.4]
  ORR per iRECIST | 16.7 [2.1 to 48.4]

6. Secondary Outcome: Phase 1b/2a: Duration of Objective Response (DOR)
Description: DOR was defined as the time from the first occurrence of a documented objective response to the time of the first documented disease progression or death from any cause, whichever occurs first, per RECIST 1.1 and iRECIST as determined by the investigator.
Time Frame: Up to 2 years
Population: Efficacy Evaluable Analysis Set: all participants who received at least one dose of both the trialmedication (NT-I7 and Pembrolizumab) and had an evaluable baseline and at least one evaluable post-baseline assessment of tumor response. Only participants who had a documented response were included.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1b: Dose Level 1 (NT-I7 480 ug/kg) | Phase 1b: Dose Level 2 (NT-I7 960 ug/kg) | Phase 1b: Dose Level 3 (NT-I7 1200 ug/kg) | Phase 2a: Arm I | Phase 2a: Arm II | Phase 2a: Arm III | Phase 2a: Arm IV | Phase 2a: Arm IVa | Phase 2a: Arm V | Phase 2a: Arm Va | Phase 2a: Biomarker Cohort
Number analyzed (Participants) | 2 | 0 | 0 | 0 | 1 | 2 | 3 | 0 | 2 | 1 | 2
months
  DOR per RECIST 1.1: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 1 | 2
  DOR per RECIST 1.1 | NA [NA to NA] — The median and/or its confidence intervals could not be estimated due to the limited number of events among responders (many participants were censored). |  |  |  |  | NA [4.2 to NA] — The median and/or its confidence intervals could not be estimated due to the limited number of events among responders (many participants were censored). | 13.1 [NA to NA] — The median and/or its confidence intervals could not be estimated due to the limited number of events among responders (many participants were censored). |  | NA [NA to NA] — The median and/or its confidence intervals could not be estimated due to the limited number of events among responders (many participants were censored). | 8.6 [NA to NA] — The median and/or its confidence intervals could not be estimated due to the limited number of events among responders (many participants were censored). | NA [7.0 to NA] — The median and/or its confidence intervals could not be estimated due to the limited number of events among responders (many participants were censored).
  DOR per iRECIST | NA [NA to NA] — The median and/or its confidence intervals could not be estimated due to the limited number of events among responders (many participants were censored). |  |  |  | 4.8 [NA to NA] — The median and/or its confidence intervals could not be estimated due to the limited number of events among responders (many participants were censored). | NA [4.2 to NA] — The median and/or its confidence intervals could not be estimated due to the limited number of events among responders (many participants were censored). | 13.0 [13.0 to NA] — The median and/or its confidence intervals could not be estimated due to the limited number of events among responders (many participants were censored). |  | NA [9.7 to NA] — The median and/or its confidence intervals could not be estimated due to the limited number of events among responders (many participants were censored). | 8.6 [NA to NA] — The median and/or its confidence intervals could not be estimated due to the limited number of events among responders (many participants were censored). | NA [7.0 to NA] — The median and/or its confidence intervals could not be estimated due to the limited number of events among responders (many participants were censored).

7. Secondary Outcome: Phase 1b/2a: Disease Control Rate (DCR)
Description: DCR was defined as the proportion of participants with a best overall response of CR, PR, stable disease (SD) per RECIST 1.1 and iRECIST as determined by the investigator..
  SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD) at least a 20% increase in the sum of the diameters of target lesions), taking as reference the smallest sum diameters while on study.
Time Frame: Up to 2 years
Population: Efficacy Evaluable Analysis Set: all participants who received at least one dose of both the trial medications (NT-I7 and Pembrolizumab) and had an evaluable baseline and at least one evaluable post-baseline assessment of tumor response.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1b: Dose Level 1 (NT-I7 480 ug/kg) | Phase 1b: Dose Level 2 (NT-I7 960 ug/kg) | Phase 1b: Dose Level 3 (NT-I7 1200 ug/kg) | Phase 2a: Arm I | Phase 2a: Arm II | Phase 2a: Arm III | Phase 2a: Arm IV | Phase 2a: Arm IVa | Phase 2a: Arm V | Phase 2a: Arm Va | Phase 2a: Biomarker Cohort
Number analyzed (Participants) | 3 | 3 | 6 | 14 | 26 | 15 | 27 | 26 | 26 | 26 | 12
percentage of participants
  DCR per RECIST 1.1 | 66.7 [9.4 to 99.2] | 0 [0.0 to 70.8] | 66.7 [22.3 to 95.7] | 21.4 [4.7 to 50.8] | 42.3 [23.4 to 63.1] | 20.0 [4.3 to 48.1] | 40.7 [22.4 to 61.2] | 30.8 [14.3 to 51.8] | 30.8 [14.3 to 51.8] | 19.2 [6.6 to 39.4] | 25.0 [5.5 to 57.2]
  DCR per iRECIST | 66.7 [9.4 to 99.2] | 0 [0.0 to 70.8] | 66.7 [22.3 to 95.7] | 21.4 [4.7 to 50.8] | 50.0 [29.9 to 70.1] | 20.0 [4.3 to 48.1] | 44.4 [25.5 to 64.7] | 34.6 [17.2 to 55.7] | 34.6 [17.2 to 55.7] | 19.2 [6.6 to 39.4] | 25.0 [5.5 to 57.2]

8. Secondary Outcome: Phase 1b/2a: Progression Free Survival (PFS)
Description: PFS was defined as the time from the first trial treatment (Cycle 1, Day 1) to the first occurrence of progression or death from any cause, whichever occurs first per RECIST 1.1 and iRECIST as determined by the investigator.
  PD was defined as at least a 20% increase in the sum of the diameters of target lesions, using the smallest sum observed on study as reference, with an absolute increase of at least 5 mm, or the appearance of new lesions, or unequivocal progression of non-target lesions, per RECIST 1.1.
Time Frame: Up to 2 years
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Pase 2a: Arm IV: CPI naïve participants with R/R MSS-CRC received NT-I7 at the RP2D (1200 ug/kg) as an IM injection Q6W, on Day 1 of alternate cycles (Cycle 1, 3, 5 etc.). Participants received 200 mg Pembrolizumab as an IV infusion Q3W, on Day 1 of every cycle (cycle duration= 21 days).
Arm/Group | Phase 1b: Dose Level 1 (NT-I7 480 ug/kg) | Phase 1b: Dose Level 2 (NT-I7 960 ug/kg) | Phase 1b: Dose Level 3 (NT-I7 1200 ug/kg) | Phase 2a: Arm I | Phase 2a: Arm II | Phase 2a: Arm III | Pase 2a: Arm IV | Phase 2a: Arm IVa | Phase 2a: Arm V | Phase 2a: Arm Va | Phase 2a: Biomarker Cohort
Number analyzed (Participants) | 3 | 3 | 6 | 14 | 26 | 15 | 27 | 26 | 26 | 26 | 12
months
  PFS per RECIST 1.1 | 8.6 [1.1 to NA] — The median and/or its confidence interval could not be estimated due to the limited number of events. | 1.3 [0.9 to NA] — The median and/or its confidence interval could not be estimated due to the limited number of events. | 5.3 [1.2 to NA] — The median and/or its confidence interval could not be estimated due to the limited number of events. | 1.2 [1.0 to 1.3] | 1.4 [1.3 to 4.1] | 1.3 [1.2 to 1.4] | 1.7 [1.4 to 2.7] | 1.4 [1.4 to 1.9] | 1.4 [1.3 to 1.4] | 1.3 [1.2 to 1.3] | 1.4 [1.2 to 1.4]
  PFS per iRECIST | NA [1.1 to NA] — The median and/or its confidence interval could not be estimated due to the limited number of events. | NA [1.3 to NA] — The median and/or its confidence interval could not be estimated due to the limited number of events. | NA [1.4 to NA] — The median and/or its confidence interval could not be estimated due to the limited number of events. | 3.8 [1.3 to NA] — The median and/or its confidence interval could not be estimated due to the limited number of events. | 4.1 [1.4 to NA] — The median and/or its confidence interval could not be estimated due to the limited number of events. | 4.0 [1.6 to 11.4] | 2.7 [1.7 to NA] — The median and/or its confidence interval could not be estimated due to the limited number of events. | 7.9 [2.4 to NA] — The median and/or its confidence interval could not be estimated due to the limited number of events. | 4.4 [1.5 to NA] — The median and/or its confidence interval could not be estimated due to the limited number of events. | 1.3 [1.3 to 2.1] | 4.1 [1.3 to NA] — The median and/or its confidence interval could not be estimated due to the limited number of events.

9. Secondary Outcome: Phase 1b/2a: Overall Survival (OS)
Description: OS was defined as the time from first trial treatment (Cycle 1, Day 1) to death from any cause.
Time Frame: Up to 2 years
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Phase 2a: Arm I: CPI treated participants with R/R TNBC received NT-I7 at RP2D (1200 ug/kg) as an IM injection Q6W, on Day 1 of alternate cycles (Cycle 1, 3, 5 etc.). Participants received 200 mg Pembrolizumab as an IV infusion Q3W, on Day 1 of every cycle (cycle duration= 21 days).
Arm/Group | Phase 1b: Dose Level 1 (NT-I7 480 ug/kg) | Phase 1b: Dose Level 2 (NT-I7 960 ug/kg) | Phase 1b: Dose Level 3 (NT-I7 1200 ug/kg) | Phase 2a: Arm I | Phase 2a: Arm II | Phase 2a: Arm III | Phase 2a: Arm IV | Phase 2a: Arm IVa | Phase 2a: Arm V | Phase 2a: Arm Va | Phase 2a: Biomarker Cohort
Number analyzed (Participants) | 3 | 3 | 6 | 14 | 26 | 15 | 27 | 26 | 26 | 26 | 12
months | NA [19.2 to NA] — The median and/or its confidence interval could not be estimated due to the limited number of events. | 9.4 [NA to NA] — The median and/or its confidence interval could not be estimated due to the limited number of events. | NA [14.0 to NA] — The median and/or its confidence interval could not be estimated due to the limited number of events. | 9.1 [3.8 to 10.3] | 17.3 [10.5 to 31.0] | 5.9 [2.1 to 16.3] | 9.3 [7.8 to 18.5] | 16.0 [7.1 to 24.0] | 11.1 [3.6 to 26.2] | 6.7 [2.9 to 10.9] | 10.1 [3.7 to 22.9]

10. Secondary Outcome: Phase 1b/2a: Number of Participants Who Experienced an Increase in Anti-Drug Antibodies (ADAs) to NT-I7
Description: Immunogenicity to NT-I7 was measured using a risk-based, tiered testing approach. This included screening and confirmatory assays for binding ADAs, epitope-specific assays to characterize ADA reactivity to whole NT-I7 vs IL-7 domain, and a cell-based neutralizing ADA assay for IL7 bioactivity. Participants' samples were obtained at baseline and over the course of treatment (to evaluate the prevalence and incidence of treatment-emergent/boosted ADA).
  Not detected or detected but not confirmed ADA was defined as negative. Detected and confirmed ADA was defined as positive.
Time Frame: Up to 2 years
Population: Safety Analysis Set: all participants who received at least one dose (even partially) of one or both trial medications.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Dose Level 1 (NT-I7 480 ug/kg) | Phase 1b: Dose Level 2 (NT-I7 960 ug/kg) | Phase 1b: Dose Level 3 (NT-I7 1200 ug/kg) | Phase 2a: Arm I | Phase 2a: Arm II | Phase 2a: Arm III | Phase 2a: Arm IV | Phase 2a: Arm IVa | Phase 2a: Arm V | Phase 2a: Arm Va | Phase 2a: Biomarker Cohort
Number analyzed (Participants) | 3 | 3 | 6 | 16 | 34 | 17 | 29 | 28 | 32 | 34 | 13
Participants
  Participants with ADA positive at baseline | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 1 | 0
  Participants with post-dose ADA positive | 3 | 1 | 6 | 3 | 24 | 0 | 22 | 19 | 27 | 14 | 2

11. Secondary Outcome: Biomarker Cohort: Number of Participants Who Experienced TEAEs, SAEs, Trial Treatment-related TEAEs and Trial Treatment-related SAEs
Description: A TEAE was any AE that starts on/after the first day of trial treatment or that worsens on/after the first day of trial treatment and up to 30 days (90 days for serious adverse events) after the date of last dose of trial drugs, or initiation of new anticancer therapy, whichever is earlier. A SAE was defined as any AE that resulted in any of the following outcomes:
  Death; A life-threatening AE; An AE that resulted in inpatient hospitalization or prolongation of existing hospitalization for ≥24 hours; A persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions; A congenital anomaly/birth defect; Important Medical Events (IME) that may not result in death, be life threatening, or require hospitalization may be considered serious when, based upon medical judgment, they may jeopardize the participant and may require medical or surgical intervention to prevent one of the outcomes listed in this definition.
Time Frame: Up to 2 years and 3 months
Population: Safety Analysis Set: all participants who received at least one dose (even partially) of one or both trial medications. Only participants in the Biomarker Cohort were analyzed for this Outcome Measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2a: Biomarker Cohort
Number analyzed (Participants) | 13
Participants
  TEAEs | 13
  SAEs | 9
  Trial Treatment-related TEAEs | 10
  Trial Treatment-related SAEs | 0

ADVERSE EVENTS:
Time Frame: Up to 2 years and 3 months
Description: A TEAE was any AE that starts on/after the first day of trial treatment or that worsens on/after the first day of trial treatment and up to 30 days (90 days for serious adverse events) after the date of last dose of trial drugs, or initiation of new anticancer therapy, whichever is earlier.
  Safety Analysis Set: all participants who received at least one dose (even partially) of one or both trial medications. For Biomarker Cohort: AEs in this arm were reported as a whole, not by dose level.
Arm/Group | Phase 1b: Dose Level 1 (NT-I7 480 ug/kg) | Phase 1b: Dose Level 2 (NT-I7 960 ug/kg) | Phase 1b: Dose Level 3 (NT-I7 1200 ug/kg) | Phase 2a: Arm I | Phase 2a: Arm II | Phase 2a: Arm III | Phase 2a: Arm IV | Phase 2a: Arm IVa | Phase 2a: Arm V | Phase 2a: Arm Va | Phase 2a: Biomarker Cohort
All-Cause Mortality (participants affected / at risk) | 1/3 | 1/3 | 1/6 | 9/16 | 20/34 | 12/17 | 19/29 | 16/28 | 18/32 | 24/34 | 8/13
Serious Adverse Events (participants affected / at risk) | 2/3 | 1/3 | 1/6 | 4/16 | 28/34 | 11/17 | 15/29 | 20/28 | 18/32 | 27/34 | 9/13
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 6/6 | 16/16 | 34/34 | 17/17 | 29/29 | 27/28 | 32/32 | 34/34 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b: Dose Level 1 (NT-I7 480 ug/kg) (N=3) | Phase 1b: Dose Level 2 (NT-I7 960 ug/kg) (N=3) | Phase 1b: Dose Level 3 (NT-I7 1200 ug/kg) (N=6) | Phase 2a: Arm I (N=16) | Phase 2a: Arm II (N=34) | Phase 2a: Arm III (N=17) | Phase 2a: Arm IV (N=29) | Phase 2a: Arm IVa (N=28) | Phase 2a: Arm V (N=32) | Phase 2a: Arm Va (N=34) | Phase 2a: Biomarker Cohort (N=13)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 4 | 0 | 3
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Obstruction gastric (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Duodenal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Immune-mediated gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Malignant ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rectal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 7 | 4 | 3 | 4 | 5 | 14 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Extradural neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 2 | 0 | 4 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Malignant pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 9 | 0 | 1 | 1 | 0 | 2 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 1 | 3 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Abdominal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Biliary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Peritonitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rectal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Spontaneous bacterial peritonitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 2 | 3 | 2
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Immune-mediated nephritis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 2 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
SJS-TEN overlap (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Jugular vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Immune thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Myocarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cholangitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Addisons disease (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vitreous haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b: Dose Level 1 (NT-I7 480 ug/kg) (N=3) | Phase 1b: Dose Level 2 (NT-I7 960 ug/kg) (N=3) | Phase 1b: Dose Level 3 (NT-I7 1200 ug/kg) (N=6) | Phase 2a: Arm I (N=16) | Phase 2a: Arm II (N=34) | Phase 2a: Arm III (N=17) | Phase 2a: Arm IV (N=29) | Phase 2a: Arm IVa (N=28) | Phase 2a: Arm V (N=32) | Phase 2a: Arm Va (N=34) | Phase 2a: Biomarker Cohort (N=13)
Fatigue (General disorders) | 1 | 0 | 4 | 4 | 14 | 8 | 13 | 12 | 12 | 16 | 4
Pyrexia (General disorders) | 3 | 0 | 3 | 5 | 5 | 1 | 12 | 12 | 14 | 9 | 2
Injection site reaction (General disorders) | 2 | 1 | 0 | 2 | 5 | 3 | 9 | 9 | 7 | 7 | 4
Oedema peripheral (General disorders) | 1 | 2 | 2 | 5 | 8 | 2 | 7 | 2 | 5 | 9 | 3
Chills (General disorders) | 2 | 0 | 5 | 2 | 2 | 0 | 5 | 2 | 7 | 1 | 1
Influenza like illness (General disorders) | 0 | 0 | 1 | 3 | 3 | 1 | 5 | 4 | 3 | 4 | 1
Injection site pain (General disorders) | 0 | 0 | 4 | 2 | 6 | 2 | 2 | 2 | 2 | 0 | 1
Injection site erythema (General disorders) | 0 | 0 | 4 | 0 | 4 | 2 | 1 | 1 | 2 | 2 | 1
Injection site pruritus (General disorders) | 0 | 0 | 2 | 2 | 3 | 2 | 1 | 1 | 2 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 1 | 1 | 0 | 0
Injection site oedema (General disorders) | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0
Injection site rash (General disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 0 | 0 | 0
Injection site warmth (General disorders) | 0 | 0 | 2 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 2 | 0
Injection site induration (General disorders) | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1
Early satiety (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Generalised oedema (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Axillary pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Injection site nodule (General disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Device related thrombosis (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hernia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injection site bruising (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Injection site dryness (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Performance status decreased (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaccination site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 3 | 4 | 10 | 1 | 14 | 3 | 10 | 5 | 2
Vomiting (Gastrointestinal disorders) | 2 | 0 | 1 | 2 | 8 | 1 | 12 | 3 | 6 | 2 | 1
Constipation (Gastrointestinal disorders) | 2 | 0 | 2 | 2 | 5 | 2 | 2 | 7 | 6 | 7 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 5 | 1 | 9 | 5 | 7 | 4 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 2 | 2 | 5 | 3 | 5 | 3 | 4 | 4 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 6 | 3 | 3
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 4 | 2 | 4 | 2 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 2 | 4 | 2 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Oral dysaesthesia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Malignant ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal mass (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fistula of small intestine (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lip oedema (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mucous stools (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oral mucosal blistering (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pancreatic failure (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 2 | 2 | 6 | 6 | 4 | 10 | 8 | 9 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 3 | 1 | 7 | 3 | 8 | 7 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 4 | 4 | 2 | 5 | 4 | 3 | 6 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 3 | 2 | 6 | 2 | 6 | 4 | 1 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 4 | 3 | 4 | 7 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2 | 3 | 1 | 4 | 4 | 2 | 4 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 4 | 1 | 3 | 2 | 4 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 3 | 3 | 2 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 4 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 1 | 2 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 1 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 2
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Appetite disorder (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 2 | 8 | 4 | 7 | 8 | 8 | 3 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 4 | 6 | 1 | 8 | 6 | 7 | 7 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 4 | 5 | 3 | 1 | 4 | 8 | 8 | 4
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 2 | 1 | 1 | 1 | 2 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 2 | 2 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypohidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pruritus allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin hypertrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 3 | 1 | 1 | 3 | 5 | 7 | 5 | 5
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 5 | 1 | 3 | 3 | 4 | 3 | 7 | 1
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 3 | 3 | 1 | 5 | 4 | 5 | 5 | 0
Weight decreased (Investigations) | 0 | 0 | 1 | 1 | 6 | 3 | 4 | 3 | 3 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 2 | 3 | 2 | 6 | 6 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 2 | 6 | 2 | 5 | 2 | 3
Platelet count decreased (Investigations) | 0 | 0 | 1 | 1 | 0 | 2 | 1 | 4 | 2 | 3 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 1 | 0 | 1 | 0 | 3 | 1 | 2 | 3 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 5 | 0 | 3
Weight increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 2 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 1 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 2 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1
Lymphocyte count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Breath sounds abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Blood cholesterol increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood iron decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oxygen saturation decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Prothrombin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Right ventricular systolic pressure increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urine analysis abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 3 | 4 | 3 | 7 | 3 | 5 | 6 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 5 | 5 | 2 | 6 | 5 | 3 | 3 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 3 | 2 | 0 | 3 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 1 | 0 | 3 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 1 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 2 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 3 | 0 | 0 | 1 | 0
Malignant pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 2 | 1 | 2 | 4 | 3 | 5 | 4 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3 | 1 | 0 | 1 | 3 | 2 | 3 | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 3 | 1 | 1 | 4 | 2 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 3 | 2 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2 | 2 | 0 | 2 | 1 | 1 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 0 | 2 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Immune-mediated arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Autoimmune arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Spinal deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 3 | 0 | 0 | 1 | 6 | 1 | 5 | 3 | 1 | 4 | 2
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 2 | 2 | 3 | 2 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 3 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 1 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Taste disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Horners syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Psychomotor hyperactivity (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vasogenic cerebral oedema (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vocal cord paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 2 | 3 | 1 | 6 | 6 | 6 | 11 | 4
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 2
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Immune thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Splenic vein thrombosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 1 | 1 | 3 | 2 | 2 | 6 | 0 | 2 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 6 | 0 | 2 | 0 | 1 | 4 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 3 | 1 | 0 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abscess oral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Epstein-Barr virus infection reactivation (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Klebsiella urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Liver abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lymph gland infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rectal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 2 | 0 | 0 | 0 | 7 | 1 | 4 | 2 | 5 | 2 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 2 | 2 | 1 | 2 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Cyanosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Embolism venous (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vena cava embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vena cava thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 0 | 0 | 1 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 2 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 2
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Bladder dilatation (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bladder hypertrophy (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bladder obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal vein thrombosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary hesitation (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urine flow decreased (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 2 | 3 | 3 | 1 | 1 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 1 | 3 | 1 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Immunisation reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasal injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Spinal column injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 5 | 3 | 1 | 3 | 1
Tachycardia (Cardiac disorders) | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 3 | 1 | 3 | 2 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 2 | 0 | 2 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Hallucination, visual (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Libido decreased (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 5 | 2 | 4 | 3 | 2
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypercalcaemia of malignancy (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thyroiditis (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 1
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Eye swelling (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Macular oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Retinal vein occlusion (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vitreous haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tumour thrombosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Perineal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Deafness unilateral (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Motion sickness (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bile duct stenosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hepatic vein thrombosis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-10-26): https://cdn.clinicaltrials.gov/large-docs/53/NCT04332653/Prot_000.pdf
  • Statistical Analysis Plan (2025-05-01): https://cdn.clinicaltrials.gov/large-docs/53/NCT04332653/SAP_001.pdf